CLINICAL TRIAL: NCT05108376
Title: Feasibility and Initial Clinical Impressions of Predictive Monitoring Integrated With the RACE Team
Acronym: VSI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 3199
Record Dates: First submitted 2021-10-07; First posted 2021-11-04 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Deterioration, Clinical
MeSH Terms: conditions — Clinical Deterioration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Arm (Experimental): The Visensia Safety Index (VSI) will be used to alert RACE staff of patient deterioration.
  Interventions: Device: Visensia Safety Index (VSI)

INTERVENTIONS:
Device: Visensia Safety Index (VSI) — Enrolled patients will undergo continuous vital sign monitoring, to be used by the Visensia Safety Index (VSI) to identify early deterioration. If early deterioration is identified, the VSI will produce an alert to notify the RACE team.

SUMMARY:
Rapid response teams (RRTs) have been adopted by hospitals to provide urgent critical care to hospitalized patients who require quick intervention to prevent further deterioration. Early warning scores (EWS) serve as a method to identify patients requiring RRT assessment by analyzing routinely collected data such as vital signs and laboratory results. The Visensia Safety Index (VSI) is an EWS that uses continuous vital sign monitoring and machine learning to identify the likelihood of deterioration and can be integrated with existing hospital data infrastructure. Initial studies of the VSI have both validated the system and found that patients monitored using VSI had a shorter duration of any instability and fewer episodes of serious and persistent instability. The investigators' recent retrospective analysis at The Ottawa Hospital (TOH) identified that implementation of an EWS could have detected earlier deterioration in over half of the patients identified, potentially preventing subsequent ICU admission, severity of illness, and/or mortality. Thus, this study aims to determine the feasibility and potential impact of implementing a portable continuous monitoring system with a VSI trigger at TOH to identify patients at high risk of deterioration.

ELIGIBILITY:
Inclusion Criteria:

Adult patient (greater than or equal to 18 years of age) designated for the most aggressive levels of potential intervention (Category 1 status - Full Care and Category 2 status - Full Care except CPR) who belong to one of the following groups:

* Patients who have undergone high risk elective surgery (Whipple procedures, high risk vascular surgery, high risk general surgery, among others)
* Malignant haematology or oncology patients at high risk for deterioration
* Patients with infection admitted from the Emergency Department (ED) to the ward
* Other high-risk patients determined at the discretion of the clinical team

Exclusion Criteria:

* Patients admitted to a unit with higher level monitoring (Neurological Acute Assessment Unit, Acute Monitoring Area, Trauma Step-Down, Intensive Care Unit)
* Patients with Category III (Full Care except Respiratory or Hemodynamic Life Support, or CPR) or IV status (Comfort Care)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate technical feasibility of collecting greater than 80% of continuous data | Upon study completion, 10 months after study initiation
  Feasibility of continuous data collection will be evaluated by determining if greater than 80% of continuous data can be collected
Evaluate technical feasibility of feeding greater then 80% of continuous data to the predictive tool | Upon study completion, 10 months after study initiation
  Feasibility of feeding continuous data to the predictive tool will evaluated by determining if greater than 80% of continuous data can be fed to the predictive tool
Evaluate technical feasibility of updating the predictive tool on a regular basis greater than 80% of the time | Upon study completion, 10 months after study initiation
  Feasibility of updating the predictive tool on a regular basis will be evaluated by determining if greater than 80% of the time the predictive tool can be updated on a regular basis
Evaluate technical feasibility of reporting greater then 80% of triggers to the RACE team | Upon study completion, 10 months after study initiation
  Feasibility of reporting triggers to the RACE team will be evaluated by determining if greater than 80% of triggers are reported to the RACE team
Evaluate clinical feasibility by assessing MD opinions of the VSI | Upon study completion, 10 months after study initiation
  Clinical feasibility will be evaluated by assessing MD opinions regarding understanding of the predictive tool, ease of use, perceived strengths and limitations, and perceived enablers and barriers to effective usage through post-encounter surveys and interviews
Evaluate clinical feasibility by assessing RN opinions of the VSI | Upon study completion, 10 months after study initiation
  Clinical feasibility will be evaluated by assessing RN opinions regarding understanding of the predictive tool, ease of use, perceived strengths and limitations, and perceived enablers and barriers to effective usage through post-encounter surveys and interviews
Evaluate clinical feasibility by assessing RT opinions of the VSI | Upon study completion, 10 months after study initiation
  Clinical feasibility will be evaluated by assessing RT opinions regarding understanding of the predictive tool, ease of use, perceived strengths and limitations, and perceived enablers and barriers to effective usage through post-encounter surveys and interviews
Evaluate financial feasibility of implementing the VSI system | Upon study completion, 10 months after study initiation
  Financial feasibility of implementing the VSI system will be evaluated by identifying the costs related to implementation and maintenance of the portable continuous monitoring system through health economic evaluation

SECONDARY OUTCOMES:
Evaluate potential clinical impact of the VSI | Upon study completion, 10 months after study initiation
  The potential clinical impact of the VSI will be evaluated by comparing the prognostic accuracy of the VSI trigger to clinical gestalt using statistical analysis of performance measures including sensitivity, specificity, positive predictive value, negative predictive value, and area under the curve.
Evaluate potential financial impact of the VSI | Upon study completion, 10 months after study initiation
  The potential financial impact of the VSI will be evaluated by estimating the potential cost savings related to earlier detection of potential deterioration with comparison to historical RACE cohort

CONTACTS AND LOCATIONS:
Overall Officials: Andrew JE Seely, MD, PhD, FRCSC, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tran A, Ramchandani R, Brehaut J, Hudek N, Haines J, Watpool I, Porteous R, Kusevic D, Bucciero K, Kyeremanteng K, Hartwick M, Thavorn K, Hooper J, Kubelik D, Herry C, Scales N, Hryciw B, Abou-Khalil J, Perry J, Bredeson C, Seely A. Assessing Clinical Impressions of Early Warning Score Integration With the Rapid Response Team: Protocol for a Prospective Cohort Study. JMIR Res Protoc. 2025 Jul 31;14:e65360. doi: 10.2196/65360. PMID 40742731